CLINICAL TRIAL: NCT05262257
Title: Evaluation and Intervention of Cognitive Function in Patients With Diabetes Mellitus.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDCDstudy
Record Dates: First submitted 2021-12-28; First posted 2022-03-02 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Metformin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lifestyle intervention group (Experimental): patients did not take any hypoglycemic drugs and adopted diet, exercise and other lifestyle intervention measures to control blood sugar.
  Interventions: Behavioral: Lifestyle intervention
- Metformin treatment group (Experimental): on the basis of lifestyle intervention, patients were given metformin 2-3 times a day (starting with 2times), 0.5g each time.
  Interventions: Drug: Metformin; Behavioral: Lifestyle intervention
- Dapagliflozin treatment group (Experimental): on the basis of lifestyle intervention, patients took Dapagliflozin orally, once a day, 10mg at a time.
  Interventions: Drug: Dapagliflozin; Behavioral: Lifestyle intervention
- Healthy control group (No Intervention): no intervention.

INTERVENTIONS:
Drug: Metformin — Take it regularly for 12 weeks
  Other Names: Metformin Hydrochloride
  Arms: Metformin treatment group
Drug: Dapagliflozin — Take it regularly for 12 weeks
  Other Names: Dapagliflozin 10Mg Tab
  Arms: Dapagliflozin treatment group
Behavioral: Lifestyle intervention — patients did not take any hypoglycemic drugs and adopted diet, exercise and other lifestyle intervention measures to control blood sugar.
  Arms: Dapagliflozin treatment group; Lifestyle intervention group; Metformin treatment group

SUMMARY:
This study is a randomized controlled, single-center study of the cognitive function of diabetic patients in the Department of Endocrinology in our hospital. Through the collection of clinical data during the outpatient or hospitalization period, as well as the clinical data of follow-up at different times in the later period, the conclusion is drawn after statistical analysis. For the population who passed the observational study in the first part, patients who meet the conditions of intervention will be further screened to enter the intervention study in the second part. Patients with type 2 diabetes who meet the enrollment criteria and enter the second part are randomly divided into 3 groups according to 1:1:1; 1.Lifestyle intervention group; 2. Metformin treatment group; 3. Dapagliflozin treatment group; There are four groups with healthy control (no intervention). Follow-up review and blood samples were taken after 12 weeks respectively. After the first follow-up, follow-up can be extended to 24 weeks depending on the patient's wishes. Combined with the number of patients with diabetes in endocrinology department of our hospital in the past, and considering the nature of this study and other factors, 90 patients with type 2 diabetes and 30 healthy controls were included for research and analysis.

DETAILED DESCRIPTION:
A large amount of evidence indicates that diabetes (DM) is related to mild cognitive impairment (MCI), vascular dementia and Alzheimer disease (AD). Biological, clinical and epidemiological data all support the close link between diabetes and Alzheimer disease. AD and type 2 diabetes (T2DM) have common pathological features, including inflammation, changes in insulin signaling, or vascular damage. Event-related potential (ERP) is a specific stimulus that acts on the sensory system or a certain part of the brain. When the stimulation is given or withdrawn, the potential change in the brain area is caused. It is suitable for the assessment of brain dysfunction, especially for the assessment of people with early subclinical disease states. Among them, P300 belongs to a kind of ERP, which is an endogenous special evoked potential related to cognitive function. It can identify and evaluate early changes in cognitive function. Therefore, it can be recognized in clinical neurological or psychiatric diseases. The change of cognitive function provides reliable objective indicators, which is of great significance for early drug intervention and treatment and improving the long-term quality of life of patients. Studies have found that anti-diabetic drugs can improve cognitive and memory impairment, and have a positive effect on mitochondrial and synaptic function, neuroinflammation and brain metabolism. Anti-diabetic drugs can be developed as the treatment of MCI and AD diseases in diabetic and non-diabetic patients. Both basic and clinical trials have evidence that metformin has considerable potential for the treatment of cognitive dysfunction in T2DM. Basic experiments have confirmed that SGLT-2 inhibitors may improve the pathological state of AD, but the clinical evidence is still unclear. As the representative drug of SGLT-2, dapagliflozin, as the intervention drug in this study, focuses on its effect on improving the cognitive function of diabetic patients, and compares its effectiveness in improving cognitive function with metformin.

This study is a randomized controlled, single-center study of the cognitive function of diabetic patients in the Department of Endocrinology in our hospital. Through the collection of clinical data during the outpatient or hospitalization period, as well as the clinical data of follow-up at different times in the later period, the conclusion is drawn after statistical analysis. For the population who passed the observational study in the first part, patients who meet the conditions of intervention will be further screened to enter the intervention study in the second part. Patients with type 2 diabetes who meet the enrollment criteria and enter the second part are randomly divided into 3 groups according to 1:1:1;1.Lifestyle intervention group; 2. Metformin treatment group; 3. Dapagliflozin treatment group; There are four groups with healthy control (no intervention). Follow-up review and blood samples were taken after 12 weeks respectively. After the first follow-up, follow-up can be extended to 24 weeks depending on the patient's wishes. Combined with the number of patients with diabetes in endocrinology department of our hospital in the past, and considering the nature of this study and other factors, 90 patients with type 2 diabetes and 30 healthy controls were included for research and analysis.

ELIGIBILITY:
Inclusion Criteria:

1. some patients with type 2 diabetes were observed and studied:

   * type 2 diabetes was diagnosed according to the 1999 WHO standard and the course of disease was less than 1 year;
   * no hypoglycemic drugs were used or stopped for more than 12 weeks;
   * 40-60 years old (including both ends);
   * able to understand the procedures and methods of this study, willing to strictly abide by the clinical trial plan to complete the trial, and voluntarily signed the informed consent form.
2. healthy controls were age, sex and weight matching:

   * 40-60 years old (including both ends);
   * normal blood glucose: fasting blood glucose<6.1mmol/l, postprandial 2-hour blood glucose <7.8mmol /l;
   * able to understand the procedures and methods of this study, willing to strictly abide by the clinical trial plan to complete this trial, and voluntarily signed the informed consent form.

Exclusion Criteria:

* pregnancy or lactation;
* acute complications (including DKA, hypertonic coma) not corrected;
* history of cerebral hemorrhage and stroke;
* other neurological and mental disorders that clearly affect cognitive function, such as anxiety, depression, AD, PD;
* the New York Heart Association (NYHA) defines congestive heart failure as Class III or IV;
* active liver disease and / or obvious abnormal liver function, defined as AST >2.5 times the normal upper limit and / or ALT>2.5 times the normal upper limit and / or total bilirubin > 1.5 times the normal upper limit;
* moderate and severe renal insufficiency [using CKD-EPI formula to calculate eGFR<60ml/ (min*1.73m2)];
* malignant tumor has not been cured;
* AD family history (first-degree relatives such as parents, siblings, children, etc.). (10) Alcohol or drug abuse within 3 months, which, according to the researchers, may affect the participants' participation in the study or the status of the subjects, resulting in drug use or compliance during the trial (alcohol abuse is defined as alcohol intake of more than 15g a day for women and more than 25g for men (15g alcohol equals 450mL beer, 150mL wine or 50mL low spirits), more than twice a week);
* long-term intravenous administration, oral administration and intra-articular administration of corticosteroids for more than 7 days within 2 months before screening;
* patients with thyroid dysfunction with unstable treatment dose within 3 months (such as thiourea, thyroid hormones);
* severe trauma or infection that may affect blood glucose control within 1 month;
* patients with severe systemic diseases who were judged by the researchers to be unsuitable for enrollment;
* conditions that other researchers considered inappropriate to participate in this clinical trial.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Event-related potential (ERP) | 12 weeks
  Event-related potential (ERP) is a potential change in a region of the brain caused by the addition of a specific stimulus to a specific part of the sensory system or brain when the stimulus is given or withdrawn. It is suitable for the assessment of cerebral dysfunction, especially for the population with early subclinical disease. Among them, P300 belongs to a kind of ERP, which is an endogenous special evoked potential related to cognitive function, and can recognize and evaluate the early changes of cognitive function, it can provide reliable and objective indexes for the change of cognitive function in clinical nerve or mental disease, and is of great significance for early drug intervention and improvement of patients'long-term quality of life.
  The measurements of P300 include the determination of the latency and amplitude of N2, P3a and P3b.
Montreal Cognitive Assessment(MoCA) | 12 weeks
  The Montreal Cognitive Assessment(MoCA) is a rapid screening tool for mild cognitive impairment (MCI) developed by Professor Nasreddine in 2004, the cognitive areas assessed included attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation and orientation. The total score of the scale was 30. The test result showed that the normal score was ≥26.
Mini-Mental State Examination(MMSE) | 12 weeks
  Mini-Mental State Examination(MMSE) includes the following seven aspects: time orientation, place orientation, immediate memory, attention and calculation, delayed memory, language, visual space. A total of 30 questions, the correct answer to each score of 1, wrong answer or do not know the score of 0, the total score of the scale ranges from 0 to 30. The test scores are closely related to the educational level, and the normal cut-off points are as follows: illiteracy>17 points, primary school>20 points, junior middle school and above>24 points.

SECONDARY OUTCOMES:
glycated hemoglobin(HbA1c、GHb) | 12 weeks
  The concentration of glycosylated hemoglobin can effectively reflect the average blood glucose level in the past 8-12 weeks. After 12 weeks of intervention, the changes of glycosylated hemoglobin in patients with type 2 diabetes reflect the therapeutic effect, and the intervention measures are adjusted according to glycosylated hemoglobin.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong KL, Chen F, Hong H, Ke X, Lv YG, Tang SS, Zhu YB. New views and possibilities of antidiabetic drugs in treating and/or preventing mild cognitive impairment and Alzheimer's Disease. Metab Brain Dis. 2018 Aug;33(4):1009-1018. doi: 10.1007/s11011-018-0227-1. Epub 2018 Apr 6. PMID 29626315
- [Background] Xue M, Xu W, Ou YN, Cao XP, Tan MS, Tan L, Yu JT. Diabetes mellitus and risks of cognitive impairment and dementia: A systematic review and meta-analysis of 144 prospective studies. Ageing Res Rev. 2019 Nov;55:100944. doi: 10.1016/j.arr.2019.100944. Epub 2019 Aug 17. PMID 31430566
- [Background] Zheng F, Yan L, Yang Z, Zhong B, Xie W. HbA1c, diabetes and cognitive decline: the English Longitudinal Study of Ageing. Diabetologia. 2018 Apr;61(4):839-848. doi: 10.1007/s00125-017-4541-7. Epub 2018 Jan 25. PMID 29368156
- [Background] Baglietto-Vargas D, Shi J, Yaeger DM, Ager R, LaFerla FM. Diabetes and Alzheimer's disease crosstalk. Neurosci Biobehav Rev. 2016 May;64:272-87. doi: 10.1016/j.neubiorev.2016.03.005. Epub 2016 Mar 9. PMID 26969101
- [Background] Cooper C, Sommerlad A, Lyketsos CG, Livingston G. Modifiable predictors of dementia in mild cognitive impairment: a systematic review and meta-analysis. Am J Psychiatry. 2015 Apr;172(4):323-34. doi: 10.1176/appi.ajp.2014.14070878. Epub 2015 Feb 20. PMID 25698435
- [Background] Patrone C, Eriksson O, Lindholm D. Diabetes drugs and neurological disorders: new views and therapeutic possibilities. Lancet Diabetes Endocrinol. 2014 Mar;2(3):256-62. doi: 10.1016/S2213-8587(13)70125-6. Epub 2013 Nov 22. PMID 24622756
- [Background] Paitel ER, Samii MR, Nielson KA. A systematic review of cognitive event-related potentials in mild cognitive impairment and Alzheimer's disease. Behav Brain Res. 2021 Jan 1;396:112904. doi: 10.1016/j.bbr.2020.112904. Epub 2020 Sep 15. PMID 32941881
- [Background] Alvarenga Kde F, Duarte JL, Silva DP, Agostinho-Pesse RS, Negrato CA, Costa OA. Cognitive P300 potential in subjects with Diabetes Mellitus. Braz J Otorhinolaryngol. 2005 Mar-Apr;71(2):202-7. doi: 10.1016/s1808-8694(15)31311-2. Epub 2005 Aug 2. PMID 16446918
- [Background] Lin B, Koibuchi N, Hasegawa Y, Sueta D, Toyama K, Uekawa K, Ma M, Nakagawa T, Kusaka H, Kim-Mitsuyama S. Glycemic control with empagliflozin, a novel selective SGLT2 inhibitor, ameliorates cardiovascular injury and cognitive dysfunction in obese and type 2 diabetic mice. Cardiovasc Diabetol. 2014 Oct 26;13:148. doi: 10.1186/s12933-014-0148-1. PMID 25344694
- [Background] Nguyen T, Wen S, Gong M, Yuan X, Xu D, Wang C, Jin J, Zhou L. Dapagliflozin Activates Neurons in the Central Nervous System and Regulates Cardiovascular Activity by Inhibiting SGLT-2 in Mice. Diabetes Metab Syndr Obes. 2020 Aug 5;13:2781-2799. doi: 10.2147/DMSO.S258593. eCollection 2020. PMID 32848437
- [Background] Wen S, Nguyen T, Gong M, Yuan X, Wang C, Jin J, Zhou L. An Overview of Similarities and Differences in Metabolic Actions and Effects of Central Nervous System Between Glucagon-Like Peptide-1 Receptor Agonists (GLP-1RAs) and Sodium Glucose Co-Transporter-2 Inhibitors (SGLT-2is). Diabetes Metab Syndr Obes. 2021 Jun 29;14:2955-2972. doi: 10.2147/DMSO.S312527. eCollection 2021. PMID 34234493
- [Background] Wicinski M, Wodkiewicz E, Gorski K, Walczak M, Malinowski B. Perspective of SGLT2 Inhibition in Treatment of Conditions Connected to Neuronal Loss: Focus on Alzheimer's Disease and Ischemia-Related Brain Injury. Pharmaceuticals (Basel). 2020 Nov 11;13(11):379. doi: 10.3390/ph13110379. PMID 33187206
- [Background] Hayden MR, Grant DG, Aroor AR, DeMarco VG. Empagliflozin Ameliorates Type 2 Diabetes-Induced Ultrastructural Remodeling of the Neurovascular Unit and Neuroglia in the Female db/db Mouse. Brain Sci. 2019 Mar 7;9(3):57. doi: 10.3390/brainsci9030057. PMID 30866531
- [Background] Fink HA, Jutkowitz E, McCarten JR, Hemmy LS, Butler M, Davila H, Ratner E, Calvert C, Barclay TR, Brasure M, Nelson VA, Kane RL. Pharmacologic Interventions to Prevent Cognitive Decline, Mild Cognitive Impairment, and Clinical Alzheimer-Type Dementia: A Systematic Review. Ann Intern Med. 2018 Jan 2;168(1):39-51. doi: 10.7326/M17-1529. Epub 2017 Dec 19. PMID 29255847
- [Background] Xu X, Sun Y, Cen X, Shan B, Zhao Q, Xie T, Wang Z, Hou T, Xue Y, Zhang M, Peng D, Sun Q, Yi C, Najafov A, Xia H. Metformin activates chaperone-mediated autophagy and improves disease pathologies in an Alzheimer disease mouse model. Protein Cell. 2021 Oct;12(10):769-787. doi: 10.1007/s13238-021-00858-3. Epub 2021 Jul 21. PMID 34291435
- [Background] Khattar D, Khaliq F, Vaney N, Madhu SV. Is Metformin-Induced Vitamin B12 Deficiency Responsible for Cognitive Decline in Type 2 Diabetes? Indian J Psychol Med. 2016 Jul-Aug;38(4):285-90. doi: 10.4103/0253-7176.185952. PMID 27570337